CLINICAL TRIAL: NCT01372228
Title: Phase I/II Pilot Study of Mixed Chimerism to Treat Inherited Metabolic Disorders
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company did not pursue this indication
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-14070-010611
Expanded Access: NCT02021266 (No longer available)
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hurler Syndrome (MPS I); Hurler-Scheie Syndrome; Hunter Syndrome (MPS II); Sanfilippo Syndrome (MPS III); Krabbe Disease (Globoid Leukodystrophy); Metachromatic Leukodystrophy (MLD); Adrenoleukodystrophy (ALD and AMN); Sandhoff Disease; Tay Sachs Disease; Pelizaeus Merzbacher (PMD); Niemann-Pick Disease; Alpha-mannosidosis
Keywords: hematopoietic stem cell Tx, chimerism, leukodystrophy
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Sudden Infant Death; Mucopolysaccharidosis III; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Adrenoleukodystrophy; Sandhoff Disease; Tay-Sachs Disease; Niemann-Pick Diseases; alpha-Mannosidosis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inherited Metabolic Disorder Patients (Experimental): Recipients are treated with hematopoietic stem cell infusion from living donors
  Interventions: Biological: hematopoietic stem cell infusion

INTERVENTIONS:
Biological: hematopoietic stem cell infusion — Enriched hematopoetic stem cell infusion

SUMMARY:
The goal of this research study is to establish chimerism and avoid graft-versus-host-disease (GVHD) in patients with inherited metabolic disorders.

DETAILED DESCRIPTION:
The objective for the study is to establish chimerism following reduced intensity conditioning with no grade III/IV GVHD. The primary endpoint we will follow is production of the missing enzyme at ≥ 10% of the normal level at day 180 post-transplant in > 90% of patients.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have a confirmed diagnosis of inherited metabolic disorder / inborn error of metabolism. Diagnosis should be confirmed by appropriate test(s) (enzyme and/or mutation analysis) before study entry. Patients must not be eligible for myeloablative chemotherapy as a preparative regimen for transplant due to age, co-morbidities or organ dysfunction.

   Inborn errors of metabolism / Inherited Metabolic Disorders (IMD) eligible for this study include the following:
   * Hurler Syndrome (MPS I)
   * Hurler-Scheie Syndrome with early neurologic involvement and/or sensitization to ERT
   * Hunter Syndrome (MPS II)
   * Sanfilippo Syndrome (MPS III)
   * Krabbe Disease (Globoid Leukodystrophy)
   * Metachromatic Leukodystrophy (MLD)
   * Adrenoleukodystrophy (ALD and AMN)
   * Sandhoff Disease
   * Tay Sachs Disease
   * Pelizaeus Merzbacher (PMD)
   * Niemann-Pick Disease
   * Alpha-mannosidosis
2. Patients must have adequate function of other organ systems as measured by:

   * Creatinine less than or equal to 2.0 mg/dl and creatinine clearance ≥60 cc/min/1.73m2. Newborns must have a creatinine clearance ≥ 25 cc/min. For babies less than or equal to 3 months of age, the raw value on glomerular filtration rate (GFR) must be ≥ 1 cc/kg/min.
   * Hepatic transaminases (ALT/AST) 2.5 x normal, bilirubin <2.0mg/dl
   * Normal cardiac function by echocardiogram or radionuclide scan (ejection fraction or shortening fraction >80% of normal value for age)
   * Pulmonary function tests (PFTs) demonstrating forced expiratory volume at one second (FEV1) of ≥50% of predicted for age. If child is too young or unable to perform PFTs, crying vital capacity result of >50% of normal value for age or resting pulse oximeter >92% on room air or clearance by pulmonologist will be required.
3. Patient must have a related donor (identical or mismatched for 1, 2 or 3 Human Leukocyte Antigen (HLA)-A, -B or -DR loci).
4. Patient, and parent, or legal guardian must have given written informed consent according to FDA guidelines.
5. Patients must have a minimum life expectancy of at least 6 months.
6. Female patients of childbearing potential cannot be pregnant or lactating/breast-feeding and must be either surgically sterile, postmenopausal (no menses for the previous 12 months), or must be practicing an effective method of birth control as determined by the investigator (e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy).
7. There is no upper or lower age limit for this study.

Exclusion Criteria

1. Patients with uncontrolled seizures, apnea, evidence of recurrent or uncontrolled aspiration, or need for chronic mechanical ventilation.
2. Patients with allogeneic stem cell transplant with cytoreductive therapy in the past 6 months.
3. Subjects must not have had previous radiation therapy that would preclude total body irradiation (TBI) (as determined by radiation therapist)
4. Uncontrolled infection or severe concomitant diseases, which in the judgment of the Principal Investigator, could not tolerate reduced intensity transplantation.
5. Subjects with a positive human immunodeficiency virus (HIV) antibody test result
6. Subjects who are pregnant, as indicated by a positive serum human chorionic gonadotropin (HCG) test
7. Subjects whose only donor is pregnant at the time of intended transplant
8. Subjects of childbearing potential who are not practicing adequate contraception as defined by the investigator at the site
9. Jehovah's witnesses being unwilling to be transfused
10. Patients that have any comorbid condition which, in the view of the Principal Investigators, renders the patient at too high a risk from treatment complications and regimen related morbidity/mortality.
11. Lack of related donors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Production of missing enzyme at levels greater than or equal to 10% of normal | Day 180 post transplant to three years

SECONDARY OUTCOMES:
Enriched Hematopoetic Stem Cell Engraftment | One month to three years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — Talaris Therapeutics Inc.
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided